CLINICAL TRIAL: NCT05898386
Title: The Effect of Education and Counseling Program Based on the Health Promotion Model on Self-Esteem, Sexual Satisfaction and Quality of Life in Women With Urinary Incontinence
Brief Title: Education and Counseling Program Based on the Health Promotion Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Esra Başkaya, Research Assistant, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-06
Record Dates: First submitted 2023-03-21; First posted 2023-06-12 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Behavior and Lifestyle Changes; Pender's Health Promotion Model; Self-Esteem; Sexual Satisfaction; Quality of Life
MeSH Terms: conditions — Urinary Incontinence; Behavior; Orgasm | interventions — Educational Status; Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention was made in the control group. The women in the control group were called during the 3-month follow-up to ask whether they received treatment for urinary incontinence simultaneously with the telephone calls of the intervention group.
- Intervention Group (Experimental): A training and counseling program based on the pender's health promotion model was applied to the intervention group.
  After the training, 3 home visits and 3 phone calls were made to support the implementation of behavioral and lifestyle changes in coping with urinary incontinence.
  Interventions: Behavioral: Behaviour and Lifestyle Changes in Urinary Incontinence

INTERVENTIONS:
Behavioral: Behaviour and Lifestyle Changes in Urinary Incontinence — The women included in the second stage were given a pre-test before the training program. Training program included behavioral and lifestyle changes in coping with urinary incontinence
  After the training program, the women applied behavior and lifestyle changes for 3 months.
  3 home visits, 3 phone calls and 3 follow-ups were made.
  Other Names: Education and counseling program based on the 'Pender's Health Promotion Model'; Behavior and lifestyle changes training and counseling program in coping with urinary incontinence
  Arms: Intervention Group

SUMMARY:
The first phase of the study was carried out to determine the prevalence and risk factors of urinary incontinence in non-menopausal women over 18 years of age registered in a Family Health Center.

The second phase of the study was carried out to examine the effects of the education and counseling program based on the 'Pender's Health Promotion Model' on women's self-esteem, sexual satisfaction and quality of life in women with urinary incontinence.

Research Questions

What is the prevalence of UI in non-menopausal women over the age of 18 who are registered with the Family Health Center? What are the risk factors for urinary incontinence?

Research Hypotheses

H1: There is a difference between the urinary incontinence severity levels of women who received and did not receive education and counseling program based on Pender's health promotion model.

H2: There is a difference between the self-esteem levels of women who received and did not receive a training and counseling program based on Pender's health promotion model.

H3: There is a difference between the sexual satisfaction levels of women who received and did not receive the training and counseling program based on Pender's health promotion model.

H4: There is a difference between the quality of life levels of women who received training and counseling programs based on Pender's health promotion model and those who did not.

In the second stage of the study, the 'Training and Counseling Program Based on Pender's Health Promotion Model' and 'Home Monitoring and Counseling Program' were applied to the intervention group, which was prepared according to Pender's Health Promotion Model.

During the three-month period, the intervention group received 3 home visits one, two and three months after the training program, and 3 phone calls 15 days after the training program and each home visit.

No intervention was made in the control group; Data collection forms were applied simultaneously with the intervention group and they were reminded that they were in the research by making a phone call.

DETAILED DESCRIPTION:
The research was carried out in two stages.

In the first phase of the study, in a cross-sectional research design, in order to determine the prevalence and risk factors of urinary incontinence in women who are over 18 years old and who are not menopausal, registered in a Family Health Center; In this study, a pretest-posttest randomized controlled experimental research design was conducted to evaluate the effect of education and counseling program based on Pender's Health Promotion Model on self-esteem, sexual satisfaction and quality of life in women with second-stage urinary incontinence.

In the first phase of the study, 1042 women over the age of 18 who were registered at the Family Health Center and who did not go through menopause were included.

In the first stage, the data; It was collected between 18 January 2021 and 31 May 2021, using the 'Questionnaire on Descriptive Characteristics', 'International Incontinence Inquiry Form' and 'Incontinence Severity Index'.

The second stage of the study continued with 46 women who met the sample selection criteria for the second stage.

After the pre-test was completed, 46 women were assigned to the intervention and control groups (M:23, F:23) by stratified block randomization and stratified according to urinary incontinence severity (mild, moderate).

In the second stage of the research, the data; Between September 24, 2021 and January 13, 2022, 'International Incontinence Inquiry Form', 'Incontinence Severity Index', 'Information Form Based on Pender's Health Promotion Model', 'Self-Esteem Sub-Scale', 'Golombok-Rust Sexual Satisfaction Scale- It was collected using the 'Female Form', 'Incontinence Quality of Life Scale', 'Self-Efficacy/Efficacy Scale'.

In the second stage of the study, the 'Training and Counseling Program Based on Pender's Health Promotion Model' and 'Home Monitoring and Counseling Program' were applied to the intervention group, which was prepared according to Pender's Health Promotion Model.

During the three-month period, the intervention group received 3 home visits one, two and three months after the training program, and 3 phone calls 15 days after the training program and each home visit.

No intervention was made in the control group; Data collection forms were applied simultaneously with the intervention group and they were reminded that they were in the research by making a phone call.

In both stages of the study, the forms and scales were filled by the women themselves, and the women were guided during this period.

Frequency, percentage and descriptive statistics for data evaluation, Shapiro-Wilk Test, Independent Samples T-Test, Repeated Measurements Anova Test, Chi-square Test of Independence, Fisher Test, Cochran-Q Test, Mann-Whitney U Test, McNemar Test, Friedman Test and Marginal Homogeneity Test were used.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Having at least primary education level,
* Not having any mental problems,
* Not being in the pregnancy period,
* No active vaginal or urinary tract infection or gynecological malignancy,
* Not having received conservative treatment for urinary incontinence in the last 6 months,
* Not having had pelvic surgery in the last 2 months,
* No pelvic organ prolapse (POP) on stage 2,
* Mild to moderate UI,
* Not having reached menopause (diagnosed with menopause or no menstruation in the last 12 months)
* Having regular sexual intercourse,
* Not using drugs that may affect UI.

Exclusion Criteria:

* Having to take medical or surgical treatment that may affect the intervention due to a problem other than urinary incontinence during the follow-up period,
* Pregnancy during the follow-up period,
* Completion of all steps of the research.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence severity | Change from Urinary Incontinence Severity at 3 months.
  'Incontinence Severity Index' was used to measure urinary incontinence severity.
  ISI was developed by Sandvik et al. (1993) in Norway to assess the severity of UI in women with UI. ISI is a simple assessment method that can be applied easily. The validity and reliability study of ISI was conducted by Hazar and Şirin (2008), Cronbach α coefficient was 0.67; validity coefficient was determined as r=0.963 and r=0.932. In this study, the Cronbach α coefficient of ISI was found to be 0.79.
  The ISI score is calculated by multiplying the score obtained from the first question with the score obtained from the second question. Although the total score varies between 1-12; If the total ISI score is between 1-2 points, it is considered as mild, between 3-6 points as moderate, between 8-9 points as severe, and if 12 points as very severe incontinence.

SECONDARY OUTCOMES:
Frequency of urinary incontinence | Change from Frequency of urinary incontinence at 3 months.
  In the evaluation, the first, second and third dimensions are scored and the fourth dimension used in determining the UI type is not scored. The first dimension is scored as 0, 1, 2, 3, 4, 5, and the highest 5 and the lowest 0 points are taken from this dimension. The second dimension is scored as 0, 2, 4, 6, and the highest 6 and the lowest 0 points are taken from this dimension. The third dimension is scored as 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and the highest 10 and the lowest 0 points are taken from this dimension.
  The ICIQ-SF total score ranges from 0 to 21; A high score from the ICIQ-SF indicates that the quality of life of the individual is highly affected, while a low score indicates that it is less affected. Çetinel et al. (2007) in their study with 5565 women stated that when the ICIQ-SF total score is 8 and above, UI is in the dimension of disturbing and affecting daily life, and they determined 8 points as the cut-off point.
Quality of Life of women with urinary incontinence | Change from Quality of Life at 3 months.
  I-QOL consists of three sub-dimensions: limitation of behavior, psychosocial influence, and social isolation. Limitation of behaviors sub-dimension 1st, 2nd, 3rd, 4th, 10th, 11th, 13th, 20th items, psychosocial impact sub-dimension 5th, 6th, 7th, 9th, 15th, 16th, 17th, 21th, 22nd items, and the social isolation sub-dimension includes 8th, 12th, 14th, 18th, and 19th items. The five-point Likert-type scale is evaluated with "a lot" (1), "a lot" (2), "moderately" (3), "a little" (4) and "not at all" (5). The calculation of the scale is based on the scores of the I-QOL total and sub-dimensions, and the sum of each item divided by the number of items. The calculated total score is converted into a scale value from 0 to 100. An increase in the total score is considered as an increase in the quality of life.
Sexual Satisfaction | Change from Sexual Satisfaction at 3 months.
  'Golombok-Rust Inventory of Sexual Satisfaction-Women Form' was used to measure Sexual Satisfaction of women with urinary incontinence. GRISS, developed by Rust and Golombok (1986), is a measurement tool that evaluates sexual functions and the quality of sexual intercourse.
  The GRDCÖ-Female form consists of 28 items and 7 sub-dimensions: frequency of sexual intercourse, communication, satisfaction, avoidance, touch, vaginismus and anorgasmia. Items in the five-point Likert-type scale are evaluated with "never", "rarely", "sometimes", "mostly", "always" options. As the score obtained from the scale increases, the deterioration in sexual functions and the quality of the relationship increases. In the calculation of the scale, the score obtained from each sub-dimension is converted into standard scores ranging from 1 to 9. Scores of 5 and above from the sub-dimensions are considered to have a sexual problem related to that sub-dimension.
Self-esteem | Change from Self-esteem at 3 months.
  . There are a total of 6 items and 10 questions in 'Self-Esteem Sub-Scale' 5 out of 10 questions are positive and 5 are negative. 1st, 2nd and 3rd questions constitute the first item, 4th and 5th questions constitute the second item, 6th question is the third item, 7th question is the fourth item, 8th question is the fifth item, and 9th and 10th questions are the sixth item. Items are evaluated with "very true", "correct", "false" and "very false" options. Each item is 1 point; The total score that can be obtained from the scale ranges from 0 to 6. For each item, "1" is given when the individual evaluates himself negatively, and "0" when he evaluates himself positively. As the score obtained from the scale increases, the self-esteem of the individual decreases. A score of 0-1 from the scale indicates a high level of self-esteem, a score of 2-4 indicates a moderate level of self-esteem, and a score of 5-6 indicates a low level of self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Başkaya, Ankara, Eryaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study data will be shared during publication